CLINICAL TRIAL: NCT00840606
Title: A Relative Bioavailability Study of 30 mg Buspirone Hydrochloride Tablets Under Fasting Conditions
Brief Title: Buspirone Hydrochloride 30mg Tablets, Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R01-654
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Buspirone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Buspirone Hydrochloride 30 mg Tablet
- 2 (Active Comparator)
  Interventions: Drug: BUSPAR® 30 mg Tablet

INTERVENTIONS:
Drug: BUSPAR® 30 mg Tablet — 1 x 30 mg, single-dose fasting
  Arms: 2
Drug: Buspirone Hydrochloride 30 mg Tablet — 1 x 30 mg, single-dose fasting
  Arms: 1

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 30 mg Buspirone Hydrochloride Tablets by TEVA Pharmaceuticals Industries, Ltd. with that of 30 mg BUSPAR® Tablets by Bristol-Myers Squibb Company following a single oral dose (1 x 30 mg tablet) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The volunteer's body mass index (BMI) is less than or equal to 30.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems.

* The screening clinical laboratory procedures will include:

  * Hematology: hematocrit, hemoglobin, RBC count, WBC count with differential, platelet count;
  * Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase.
  * HIV antibody and hepatitis B surface antigen screens;
  * Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
  * Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, and phencyclidine;
  * Serum Pregnancy Screen (female volunteers only).
* If female and:

  * of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
  * is postmenopausal for at least 1 year; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to buspirone or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who are currently using or report using tobacco products within 90 days prior to Period I dosing.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any prescription medication or nonprescription medication in the 14 days or 7 days, respectively, prior to Period I dosing with the exception of topical products without systemic absorption.
* Volunteers who have been on an abnormal diet during the 28 days prior to Period I dosing.
* Volunteers who report an intolerance or direct venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2001-12; Primary Completion 2001-12 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | Blood samples collected over 24 hour period
Bioequivalence based on AUC0-inf | Blood samples collected over 24 hour period
Bioequivalence based on AUC0-t | Blood samples collected over 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States